CLINICAL TRIAL: NCT05942833
Title: DATE Trial: Outcomes and Quality of Life in Patients With Early Versus Elective Resection in Acute Complicated and Chronic Recurrent Left-sided Diverticulitis
Brief Title: Quality of Life in Acute Complicated and Chronic Recurrent Left-sided Diverticulitis
Acronym: DATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kepler University Hospital (Other)
Collaborators: Krankenhaus Barmherzige Schwestern Linz (Other); Elisabethinen Hospital (Other); Universitätsmedizin Mannheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1203/2022
Record Dates: First submitted 2023-06-07; First posted 2023-07-12 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2024-09

CONDITIONS: Diverticulitis of Sigmoid
Keywords: Recurrent diverticulitis; Quality of life; Acute complicated Diverticulitis; Early resection; Elective resection
MeSH Terms: conditions — Diverticulitis

STUDY DESIGN:
Intervention Model Description: prospective, randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Early) (Experimental): Early left hemicolectomy immediately up to a maximum of 2 days after 7-10 days lasting initial conservative or interventional treatment (e.g: antibiotics, analgesics, drainage) and CT scan/ultrasound proven left-sided colonic diverticulitis
  Interventions: Procedure: Sigmoid resection
- Group B (Late) (Other): Elective left hemicolectomy 6 to 8 weeks after 7-10 days lasting initial conservative or interventional treatment (e.g: antibiotics, analgesics, drainage) and CT scan/ultrasound proven left-sided colonic diverticulitis
  Interventions: Procedure: Sigmoid resection

INTERVENTIONS:
Procedure: Sigmoid resection — Timing of sigmoid resection

SUMMARY:
Patients presenting in hospital with symptoms of acute diverticulitis. Acute inflammation of the left-sided colon is confirmed with CT scan or ultrasound in experienced centers and diagnosis is defined according to the "Classification of Diverticular Disease (CDD)". CDD Type 2a, 2b and 3b will be included and then randomized in two groups. Group A will get an early left hemicolectomy 7 to 10 days after admission and initial antibiotic therapy and/or drainage of the abscess. Group B is designated for an elective resection 6 to 8 weeks after dismissal at the earliest and initial conservative treatment and/or after drainage of the abscess. Six weeks after the operation patients of Group A will be asked for their present quality of life with a standardized scoring system (Gastrointestinal Quality of Life Index = GIQLI; Short-form 36 Score = SF-36 Score; Low anterior resection syndrome = LARS Score). Group B (elective resection) will be asked at their readmission prior to elective surgery is done. This survey package will be repeated again 6 to 8 weeks later in both groups. Primary endpoints will be the two GIQLI at the said examination times. Secondary endpoints will be SF-36 score, LARS-score, GIQLI-Domains, anastomosis insufficiency and other complications, mortality and length of hospital stay. Comparisons between the groups are made at the said examination times but also 6-8 weeks after the operation.

DETAILED DESCRIPTION:
Primary endpoints:

Gastrointestinal Quality of Life Index (GIQLI)

Secondary endpoints:

SF-36 score (physical and mental health summary scores), LARS score, GIQLI-domains, anastomosis insufficiency and other complications, exitus and length of hospital stay

Treatment strategy:

A patient is coming into the hospital with acute symptoms of diverticulitis. The diagnosis must then be confirmed either with ultrasound or with a CT scan. After confirmation the patient is asked to be part of the study. At that point of time the patient does not know his randomization. After the patient's approval and signed consent the patients will bei informed about the further procedure and the appointment of surgery. Questionnaires will now be filled out and antibiotical treatment starts. If necessary a radiological intervention (drainage) is performed.

Is the patient is randomized into Group A he will get early left hemicolectomy immediately up to a maximum of 2 days after 7-10 days lasting initial conservative or interventional treatment (e.g: antibiotics, analgesics, drainage). If the patient is in Group B he will receive an elective left hemicolectomy 6 to 8 weeks after 7-10 days lasting initial conservative or interventional treatment (e.g: antibiotics, analgesics, drainage).

Reassessment of the questionnaires will bei done in both groups. Group A will be asked 6-8 after surgery and again 6-8 weeks after the second reassessment.

Group B will be asked 6-8 weeks after discharge (directly before surgery) and again 6-8 weeks after surgery.

The aim of the study is to evaluate the outcome and quality of life in patients receiving early surgery versus elective resection of the left-sided colon in acute complicated diverticulitis and chronic recurrent diverticulitis with acute exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent to participate in the study
* CDD Type 2a, 2b: acute complicated left-sided diverticulitis
* CDD Type 3b: relapsing diverticulitis without complications (>2 episodes within 2 years)
* Acute presentation
* Inflammation located in the left-sided colon
* Inflammation is CT proven or ultrasound confirmed from experienced radiologists

Exclusion Criteria:

* < 18 years
* Pregnancy
* BMI > 55kg/m2
* Current colorectal carcinoma in the left-sided colon
* Oral and/or intravenous corticosteroid
* Ongoing chemotherapy
* Status post left hemicolectomy
* Patients who cannot take care of themselves at home or are unable to follow instructions
* Patients who are not fit for surgery (anesthesia, expert knowledge from specialists) and will not benefit from surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal Quality of Life Index | Up to 18 weeks
  Quality of Life

SECONDARY OUTCOMES:
SF-36 score (Short form score) | Up to 18 weeks
  physical and mental health summary scores (0-100), the higher the better
Low anterior resection syndrome score | Up to 18 weeks
  points (0-40), the lower the better
Anastomosis insufficiency | Up to 18 weeks
  yes/no
Intraoperative complication | Up to 18 weeks
  bleeding, ureter harming (yes/no)
Exitus | Up to 18 weeks
  yes/no
Length of stay (sum of days in hospital until end of study) | Up to 18 weeks
  days
Earlier readmission due to recurrence while waiting for surgery | Up to 18 weeks
  Only in Group B
Postoperative complication | Up to 18 weeks
  pneumonia, urinary tract infection (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Shamiyeh, Dr., Principal Investigator — Kepler University Hospital Linz
Locations (4):
- Austria (3):
  - Ordensklinikum Elisabethinen Linz, Linz, Austria
  - Krankenhaus Barmherzige Schwestern Linz, Linz, Upper Austria
  - Kepler University Hospital, Linz, Upper Austria
- Universitätsklinikum Mannheim, Mannheim, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No